CLINICAL TRIAL: NCT02888769
Title: Effectiveness of Text Messaging on Risk Factors Control and Medication Adherence Among Coronary Heart Disease Patients Without Diabetes in Cardiovascular Health and Texting Messaging (CHAT) Study
Brief Title: Cardiovascular Health and Texting Messaging (CHAT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201502009-1
Record Dates: First submitted 2016-08-23; First posted 2016-09-05 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Text messages; Blood pressure; Lifestyle; Risk factors
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention-Text messaging (Experimental): Patients will receive regular semi-personalized text messages for 6 months. Each participants will receive 6 text messages per week, which will be sent at random times of the day (9.00am, 12noon, 4.00pm). Non-smokers will receive two general messages, two hypertension messages, one medication adherence message and one physical activity message per week. Smokers will receive one general message, two hypertension messages, one medication adherence message, one physical activity message and one smoking cessation message per week.
  Interventions: Behavioral: Text Messaging
- Control (No Intervention): Participants in the control group will receive 2 thank-you messages per month and undertake routine clinical practice.

INTERVENTIONS:
Behavioral: Text Messaging — Patients will receive regular semi-personalized text messages for 6 months. Each participants will receive 6 text messages per week, which will be sent at random times of the day (9.00am, 12noon, 4.00pm). Non-smokers will receive two general messages, two hypertension messages, one medication adherence message and one physical activity message per week. Smokers will receive one general message, two hypertension messages, one medication adherence message, one physical activity message and one smoking cessation message per week. Prior to study commencement, a bank of 280 messages have been developed based on guidelines and behavior change theory (BCT), and have underwent multidisciplinary expert review and qualitative review process.
  Arms: Intervention-Text messaging

SUMMARY:
The study is a two-arm, parallel, randomized clinical trial. The purpose of the study is to evaluate the effectiveness of automated mobile phone text message-based intervention for secondary prevention, including lifestyles modification, medication adherence improvement and risk factors control among coronary heart disease (CHD) patients without diabetes. The participants will be randomized into intervention and control groups in a 1:1 ratio. The intervention group will receive 6 pre-designed text messages per week in addition to usual care for 6 months, while the control group will receive usual care.

DETAILED DESCRIPTION:
Objective: This study aims to evaluate the effectiveness of automated mobile phone text message-based intervention for secondary prevention, including lifestyles modification, medication adherence improvement and risk factors control among CHD patients without diabetes. We hypothesized that an intervention using mobile phone text based education and reminder can improve risk factors control and medication adherence for CHD patients.

Study design: The study is a two-arm, parallel, randomized clinical trial. Patients will be eligible if they have documented CHD defined as having history of myocardial infarction and PCI but without diabetes mellitus, have the capability of reading and sending short message, and are able to provide informed consent. Patients who do not have an active mobile phone will be excluded. The eligible participants will be allocated into intervention and control groups in a 1:1 ratio randomly. The intervention group will receive intervention of pre-designed text messages in addition to usual care, while the control group will receive usual care. All the participants will be followed up for 6 months.

Study intervention: Participants in the intervention group will receive semi-personalized text messages for 6 months as well as usual care. Non-smokers will receive two general messages, two hypertension messages, one medication adherence message and one physical activity message per week. Smokers will receive one general message, two hypertension messages, one medication adherence message, one physical activity message and one smoking cessation message per week.

Outcome measures: The primary endpoint is systolic blood pressure control. Secondary endpoints include a change in proportion of patients achieving a systolic blood pressure<140mm Hg, physical activity, medication adherence, smoking cessation, low-density lipoprotein cholesterol (LDL-C) and body mass index (BMI). Exploratory endpoints include long-term prognosis of the patients, such as death, non-fatal myocardial infarction, stroke and so on, as well as health status (SAQ and EQ-5D).

Statistical analysis: Evaluation will be carried out on an intention-to-treat basis. Values of analyzed endpoints between intervention group and control group will be compared according to the analysis plan. We'll follow a prespecified analysis plan and subgroup analysis will be conducted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Participants with coronary artery disease defined as history of myocardial infarction and percutaneous coronary intervention (PCI)
* Capability to read and send text messages

Exclusion Criteria:

* History of diabetes
* Assumed poor adherence
* Do not have an active mobile phone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure obtained in office during each interview | Baseline; 6months
  The investigators will measure the change in systolic blood pressure from baseline to 6 months.

SECONDARY OUTCOMES:
Change in proportion of patients achieving a SBP<140mm Hg | Baseline; 6months
  The investigators will measure the proportion of patients achieving a SBP<140mm Hg from baseline to 6 months.
Change in low-density lipoprotein cholesterol (LDL-C) level | Baseline; 6months
  The investigators will measure the change in LDL-C level from baseline to 6 months.
Change in body mass index (BMI) | Baseline; 6months
  The investigators will measure the change in BMI from baseline to 6 months.
Change in medication adherence | Baseline; 6months
  The investigators will measure the change in medication adherence from baseline to 6 months.
Change in level of physical activity measured via International Physical Activity Questionnaire (IPAQ) scale | Baseline; 6months
  The investigators will measure the change in IPAQ scale from baseline to 6 months.
Change in proportion of non-smokers | Baseline; 6months
  The investigators will measure the proportion of non-smokers via self report and cotinine urine strip test from baseline to 6 months. The patients who report as non-smokers with negative cotinine test result will be defined as non-smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, MD, PhD, Principal Investigator — China National Center for Cardiovascular Disease; Harlan M Krumholz, MD, SM, Principal Investigator — Yale University
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zheng X, Spatz ES, Bai X, Huo X, Ding Q, Horak P, Wu X, Guan W, Chow CK, Yan X, Sun Y, Wang X, Zhang H, Liu J, Li J, Li X, Spertus JA, Masoudi FA, Krumholz HM. Effect of Text Messaging on Risk Factor Management in Patients With Coronary Heart Disease: The CHAT Randomized Clinical Trial. Circ Cardiovasc Qual Outcomes. 2019 Apr;12(4):e005616. doi: 10.1161/CIRCOUTCOMES.119.005616. PMID 30998400
- [Derived] Huo X, Spatz ES, Ding Q, Horak P, Zheng X, Masters C, Zhang H, Irwin ML, Yan X, Guan W, Li J, Li X, Spertus JA, Masoudi FA, Krumholz HM, Jiang L. Design and rationale of the Cardiovascular Health and Text Messaging (CHAT) Study and the CHAT-Diabetes Mellitus (CHAT-DM) Study: two randomised controlled trials of text messaging to improve secondary prevention for coronary heart disease and diabetes. BMJ Open. 2017 Dec 21;7(12):e018302. doi: 10.1136/bmjopen-2017-018302. PMID 29273661